CLINICAL TRIAL: NCT06641908
Title: A Phase 1, Two-Part, Multicenter, Open-Label First in Human Study of Anti-GD2 Antibody Drug Conjugate M3554 in Participants With Advanced Solid Tumors
Brief Title: Anti-GD2 ADC M3554 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201460_0001; 2024-513687-26-00 (Other: CTIS)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
Keywords: Glioblastoma; IDH-wildtype; Soft tissue sarcomas; GD2 prevalence; targeted therapy; TOP1 inhibitor; exatecan
MeSH Terms: conditions — Glioblastoma; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation: M3554 Monotherapy (Experimental)
  Interventions: Drug: M3554

INTERVENTIONS:
Drug: M3554 — M3554 will be administered at an escalated dose until Maximum tolerated dose (MTD) and/or a safe recommended Dose is determined in participants with STS (dose escalation A) and glioblastoma and IDH wildtype (dose escalation B).

SUMMARY:
The purpose of this study is to establish the recommended doses and further evaluate the safety and preliminary antitumor activity of M3554 in participants with soft tissue sarcoma (STS) and glioblastoma, IDH-wildtype.

Study details include:

Study Duration per participant: Approximately 4 months

ELIGIBILITY:
Inclusion Criteria:

* Escalation A: participants with documented histopathological diagnosis of locally advanced or metastatic STS with unresectable disease that has progressed after at least one prior line of anthracycline-containing systemic therapy for the locally advanced/metastatic setting.
* Participants with resectable locally advanced or metastatic disease, who had surgery before study entry will be allowed in the trial if there is residual disease after surgery and if the surgery was performed at least 4 weeks before first dose of study intervention.
* Escalation B: participants with documented histopathological diagnosis of glioblastoma, IDH-wildtype, who have progressed after ONLY one prior line of therapy (including radiotherapy +/- temozolomide, depending on the O^6-methylguanine-DNA methyltransferase [MGMT] status) and relapsing at least 3 months after the end of the radiotherapy treatment.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) below or equal to 1
* Participants with adequate hematologic, hepatic and renal function as defined in protocol
* Other protocol defined inclusion criteria could apply

  * Exclusion Criteria:
* Participant has a history of malignancy other than STS or glioblastoma (depending on the escalation/expansion cohort) within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertropia, or malignancy that in the opinion of the Investigator, is considered cured with minimal risk of recurrence within 3 years).
* STS only: Participants with history of brain metastasis, leptomeningeal metastasis, or participants with spinal cord compression
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) and Adverse Events (AEs) | up to 4 months

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Plasma Concentrations of M3554 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 or Response Assessment in Neuro-oncology (RANO) 2.0 as Assessed by Investigator | Time from randomization to planned assessment at 4 months
Duration of Response (DoR) According to RECIST Version 1.1 or RANO 2.0 as Assessed by Investigator | Time from randomization to planned assessment at 4 months
Progression-free Survival (PFS) According to RECIST Version 1.1 or RANO 2.0 as Assessed by Investigator | Time from randomization to planned assessment at 4 months
Change from Baseline in Corrected QT Interval (QTc) Interval | Pre-dose on Day 1 (baseline) up to 24 hours post-dose Day 1, Day 2, Day 5, Day 8 of Cycle 1 and Cycle 3 Day 1 (each Cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (11):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York - Memorial Sloan Kettering Cancer Center (CC)- Westc, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- UZ Leuven, Leuven, Belgium
- France (4):
  - Institut Bergonié - Service d'Oncologie Médicale, Bordeaux
  - Centre Oscar Lambret - cancerologie generale, Lille
  - Centre Leon Berard - Service d'Oncologie Medicale, Lyon
  - Centre Antoine Lacassagne - Service d'Hématologie Oncologie, Nice
- National Cancer Center Hospital, Chūōku, Japan
- Universitaetsspital Zuerich - Klinik fuer Neurologie, Zurich, Switzerland
- Royal Marsden Hospital-Sutton - Dept of Oncology (Surrey), Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201460_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html